CLINICAL TRIAL: NCT00012896
Title: Improving Cancer Pain Management Using AHCPR Cancer Pain Guidelines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: Single
Other Study IDs: NRI 97-026
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Cancers, Pain
MeSH Terms: conditions — Neoplasms; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Telephone Care + Educational (AV Materials)

INTERVENTIONS:
Behavioral: Telephone Care + Educational (AV Materials)

SUMMARY:
Cancer pain is a pervasive problem for the person with cancer. Despite advances in knowledge, effective cancer management is infrequently achieved. While this problem is multi-factorial, the patient may have attitudinal barriers to effective pain management that can be ameliorated with novel interventions.

DETAILED DESCRIPTION:
Background:

Cancer pain is a pervasive problem for the person with cancer. Despite advances in knowledge, effective cancer management is infrequently achieved. While this problem is multi-factorial, the patient may have attitudinal barriers to effective pain management that can be ameliorated with novel interventions.

Objectives:

The primary objective of this study is to determine the effects of two nursing interventions on the improvement of pain management (PM), functional status (FS) and quality of life (QOL) in veterans receiving cancer care in VA ambulatory care clinics. The two interventions will utilize selected cancer pain management strategies developed as Clinical Practice Guidelines by the Agency for Health Care Policy and Research (AHCPR). This study will test the hypothesis that those veterans in the intervention arms will have lower pain intensity scores, greater pain relief and satisfaction with PM, and will have higher QOL and FS scores specifically in the areas of physical and social functioning. A secondary aim is to measure the extent that cancer PM is affected by the intervening variables of age, affect, attitudinal barriers, veteran culture, type/stage of disease, and type of cancer treatment.

Methods:

The design of this randomized trial has one between-subjects factor, GROUP, with three levels (usual care, structured education, individualized coaching), and one within-subjects factor, TIME, with two measures, pre-test and post-test. Patients with cancer pain (n=320) are randomly assigned to one of three groups after stratifications to control for the confounding variables of pain intensity and effects of cancer treatment. Those in the structured education arm view a video on cancer pain management and receive the AHCPR patient pamphlet on cancer pain management. Those subjects in the individualized coaching arm receive the same structured education as above, but also partake in four telephone coaching sessions focusing on the individual's specific pain management problems. The primary outcome variables measured after 12 weeks are: satisfaction with pain management, quality of life and functional status.

Status:

The project is in the final phase of data analysis and writing the final report. A total of 322 subjects were recruited: 289 eligible patients completed the Pre-test and 227 completed the Post-Test. Two papers are approximately 75% written. The main study paper is in the planning stage, to be completed after the final report is submitted.

ELIGIBILITY:
Inclusion Criteria:

Patients must have a medical diagnosis of cancer, be experiencing pain as a result of their cancer or cancer treatment, be receiving treatment on an out-patient basis whereas they are taking their own medications, have a life expectancy of at least 6 months, have access to a telephone, are able to read and speak English, and do not have a drug abuse history.

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn K. Douglas, DNSc RN FAAN, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States